CLINICAL TRIAL: NCT06691373
Title: Acute Effects of Static Stretching on the Knee Joint Position Sense of Soccer Players: a Crossover Randomized Controlled Trial
Brief Title: Acute Effects of Static Stretching on the Knee Joint Position Sense of Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Fernando Pessoa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: ESS/FSA - 391/23-3
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Static Stretching; Joint Position Sense; Proprioception; Knee; Soccer
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Condition (No Intervention): 5-minute rest
- Static Stretching of 30 seconds (Active Comparator): Static stretching of the quadriceps and hamstrings for 30 seconds
  Interventions: Other: Static Stretching
- Static Stretching of 90 seconds (Active Comparator): Static stretching of the quadriceps and hamstrings for 90 seconds
  Interventions: Other: Static Stretching

INTERVENTIONS:
Other: Static Stretching — Static stretching of the quadriceps and hamstrings which was performed in the dominant limb, and held in a position where the participants referred discomfort:
  * Quadriceps - participants were in the standing position, with one hand holding the back of a chair to maintain the balance, and were instructed to pull the ankle of the lower limb to be stretched, pressing the heel towards the buttocks and, at the same time, extending the thigh;
  * Hamstrings - participants were also in the standing position, with the heel resting on a chair. They were then instructed to lean the body forward keeping the spine erect and the pelvis in anteversion, to obtain a stretch over the knee and hip.
  Arms: Static Stretching of 30 seconds; Static Stretching of 90 seconds

SUMMARY:
The aim of this study was to investigate the acute effects of static stretching on the knee joint-position sense of soccer players.

DETAILED DESCRIPTION:
This crossover randomized controlled trial included male soccer players. All participants performed 3 conditions: two experimental conditions, of static stretching of the quadriceps and hamstrings muscles, for 30 or 90 seconds; and a control condition (rest). Knee joint-position sense of the dominant limb was assessed before and immediately after the conditions for the range of 45º of knee flexion by active repositioning, using a video camera. Absolute, relative and variable angular errors were calculated.

ELIGIBILITY:
Inclusion Criteria:

* male soccer players
* aged between 18 and 30 years old
* with normal knee range of motion
* without history of lower limb injuries in the last 6 months

Exclusion Criteria:

* history of knee surgery
* with cardiorespiratory, neurological or vestibular diseases
* with positive knee integrity tests (anterior drawer, posterior drawer, Lachman test and valgus and varus stress tests)
* using drugs that could affect the central nervous system, balance, or motor control (sedatives, anxiolytics, analgesics, NSAIDs, muscle relaxants, or antibiotics).

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Absolute angular error | Change from Baseline (Pre) to Immediately after interventions or control (Post)
  The absolute value of the difference between the target range and the achieved range
Relative angular error | Change from Baseline (Pre) to Immediately after interventions or control (Post)
  The arithmetic difference between the target range and the range achieved
Variable angular error | Change from Baseline (Pre) to Immediately after interventions or control (Post)
  The standard deviation of the 3 repositionings

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde Fernando Pessoa, Porto, Portugal